CLINICAL TRIAL: NCT02739542
Title: Multi-center, Randomized, Double-blinded Assessment of Tecfidera® in Extending the Time to a First Attack in Radiologically Isolated Syndrome (RIS) (ARISE)
Brief Title: Assessment of Tecfidera® in Radiologically Isolated Syndrome (RIS)
Acronym: ARISE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, Darin Okuda, PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 102014-019
Record Dates: First submitted 2016-03-16; First posted 2016-04-15 (Estimated); Results first posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Multiple Sclerosis (MS)
Keywords: Radiologically Isolated Syndrome (RIS)
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tecfidera (Active Comparator): Tecfidera (120mg by mouth twice daily for 7 days with dose escalation to 240mg by mouth twice daily)
  Interventions: Drug: Tecfidera
- Placebo (Placebo Comparator): Placebo by mouth twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tecfidera — Blinded drug wallets will be dispensed during routine study appointments in 3 month supply, so that compliance can be reconciled at follow up visits and telephone consultations, and recorded in accountability logs.
  Other Names: Dimethyl fumarate
  Arms: Tecfidera
Drug: Placebo — Blinded drug wallets will be dispensed during routine study appointments in 3 month supply, so that compliance can be reconciled at follow up visits and telephone consultations, and recorded in accountability logs.
  Arms: Placebo

SUMMARY:
The purpose of this investigation is to systematically study the efficacy of Tecfidera in those individuals who possess incidental white matter anomalies within the brain following a MRI study that is performed for a reason other than for the evaluation of MS (multiple sclerosis).

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blinded study in which approximately 90 RIS (radiologically isolated syndrome) subjects will be treated with either Tecfidera or placebo for 2 years (1:1 randomization). Study participants, along with the treating and examining physicians, will be blinded to treatment assignment. Central Clinical and Imaging Units will screen all potential study subjects for inclusion/exclusion criteria. We expect to enroll all RIS subjects within the U.S.

Following informed consent and verification of entry criteria by the core units, study participants will be randomized 1:1 to either Tecfidera (120mg by mouth twice daily for 7 days with dose escalation to 240mg by mouth twice daily) or placebo. Clinical follow-up by the treating physician will occur at weeks 0, 48, 96, 144 and/or End of Study and during or immediately following clinical exacerbations. During clinical visits, comprehensive medical history data will be obtained by the treating physician. All reported acute or progressive clinical events will be adjudicated by the Central Clinical Unit. Clinical visits due to suspected exacerbations associated with CNS (central nervous system) demyelination, and associated diagnostic studies and treatments, will be covered under the medical standard of care by third party payers. A recommendation to re-evaluate the patient within 3 months following the clinical event to assess for extent of recovery will be made. In addition to the face-to-face visits described above, study participants will be contacted over the telephone at weeks 4, 8, 36, 60, 84, 108, and 132 to assess for medical or treatment difficulties and for study medication compliance. Standardized MRI studies of the brain will be performed at weeks 0, 96, 144 or End of Study. Clinical imaging studies of the brain and/or spinal cord performed during or immediately following the onset of a clinical exacerbation will be performed at the discretion of the site PI with scan costs covered under the medical standard of care. An end of study clinical MRI of the cervical spinal cord with and without contrast will be recommended to study participants at week 96 as medical standard of care.

ELIGIBILITY:
Inclusion criteria

1. Males and females meeting 2009 RIS criteria
2. Identified RIS cases with the initial MRI demonstrating anomalies suggestive of demyelinating disease dated > 2009
3. Incidental anomalies identified on MRI of the brain or spinal cord with the primary reason for the acquired MRI resulting from an evaluation of a process other than MS
4. CNS white matter anomalies meeting the following MRI criteria:

   * Ovoid, well-circumscribed, and homogeneous foci with or without involvement of the corpus callosum
   * T2-hyperintensities measuring > 3mm2 and fulfilling 3 of 4 Barkhof-Tintoré criteria for dissemination in space
   * CNS anomalies not consistent with a vascular pattern
   * Qualitative determination that CNS anomalies have a characteristic appearance of demyelinating lesions
5. MRI anomalies do not account for clinically apparent neurological impairments in patients

Exclusion criteria

1. Women who are pregnant or nursing
2. Incomplete medical history or radiological data
3. History of remitting clinical symptoms consistent with multiple sclerosis lasting > 24 hours prior to CNS imaging revealing anomalies suggestive of MS
4. History of paroxysmal symptoms associated with MS (i.e. Lhermitte's or Uhthoff's phenomena)
5. CNS MRI anomalies are better accounted for by another disease process
6. The subject is unwilling or unable to comply with the requirements of the study protocol
7. Exposure to a disease modifying therapy for MS/RIS within the past 3 months
8. Exposure to high-dose glucocorticosteroid treatment within the past 30 days
9. Participation in other clinical trials involving treatment with a disease-modifying agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2016-03-19 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darin T Okuda, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (11):
- United States (11):
  - Keck School of Medicine - USC - Department of Neurology, Los Angeles, California
  - Johns Hopkins University - Neurology, Baltimore, Maryland
  - Mayo Clinic Department of Neurology, Rochester, Minnesota
  - Washington University Department of Neurology, St Louis, Missouri
  - Cleveland Clinic - Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - MS Clinical Care and Research Center, Dept of Neurology, Columbia University, New York, New York
  - Oklahoma Medical Research Foundation, MS Center of Excellence, Oklahoma City, Oklahoma
  - MS Treatment Center of Dallas, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Swedish Medical Center, Seattle, Washington
  - MultiCare Institute for Research and Innovation, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polman CH, Reingold SC, Edan G, Filippi M, Hartung HP, Kappos L, Lublin FD, Metz LM, McFarland HF, O'Connor PW, Sandberg-Wollheim M, Thompson AJ, Weinshenker BG, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2005 revisions to the "McDonald Criteria". Ann Neurol. 2005 Dec;58(6):840-6. doi: 10.1002/ana.20703. PMID 16283615
- [Background] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Background] Lebrun C, Bensa C, Debouverie M, De Seze J, Wiertlievski S, Brochet B, Clavelou P, Brassat D, Labauge P, Roullet E; CFSEP. Unexpected multiple sclerosis: follow-up of 30 patients with magnetic resonance imaging and clinical conversion profile. J Neurol Neurosurg Psychiatry. 2008 Feb;79(2):195-8. doi: 10.1136/jnnp.2006.108274. PMID 18202208
- [Background] Siva A, Saip S, Altintas A, Jacob A, Keegan BM, Kantarci OH. Multiple sclerosis risk in radiologically uncovered asymptomatic possible inflammatory-demyelinating disease. Mult Scler. 2009 Aug;15(8):918-27. doi: 10.1177/1352458509106214. PMID 19667020
- [Background] Lebrun C, Blanc F, Brassat D, Zephir H, de Seze J; CFSEP. Cognitive function in radiologically isolated syndrome. Mult Scler. 2010 Aug;16(8):919-25. doi: 10.1177/1352458510375707. Epub 2010 Jul 7. PMID 20610492
- [Background] De Stefano N, Stromillo ML, Rossi F, Battaglini M, Giorgio A, Portaccio E, Hakiki B, Malentacchi G, Gasperini C, Santangelo M, Bartolozzi ML, Sormani MP, Federico A, Amato MP. Improving the characterization of radiologically isolated syndrome suggestive of multiple sclerosis. PLoS One. 2011 Apr 29;6(4):e19452. doi: 10.1371/journal.pone.0019452. PMID 21559385
- [Background] Gabelic T, Radmilovic M, Posavec V, Skvorc A, Boskovic M, Adamec I, Milivojevic I, Barun B, Habek M. Differences in oligoclonal bands and visual evoked potentials in patients with radiologically and clinically isolated syndrome. Acta Neurol Belg. 2013 Mar;113(1):13-7. doi: 10.1007/s13760-012-0106-1. Epub 2012 Jun 28. PMID 22740024
- [Background] Giorgio A, Stromillo ML, Rossi F, Battaglini M, Hakiki B, Portaccio E, Federico A, Amato MP, De Stefano N. Cortical lesions in radiologically isolated syndrome. Neurology. 2011 Nov 22;77(21):1896-9. doi: 10.1212/WNL.0b013e318238ee9b. Epub 2011 Nov 9. PMID 22076541
- [Background] Lebrun C, Le Page E, Kantarci O, Siva A, Pelletier D, Okuda DT; Club Francophone de Sclerose en Plaques (CFSEP); Radiologically Isolated Syndrome Consortium (RISC) Group. Impact of pregnancy on conversion to clinically isolated syndrome in a radiologically isolated syndrome cohort. Mult Scler. 2012 Sep;18(9):1297-302. doi: 10.1177/1352458511435931. Epub 2012 Feb 2. PMID 22300971
- [Background] Okuda DT, Mowry EM, Cree BA, Crabtree EC, Goodin DS, Waubant E, Pelletier D. Asymptomatic spinal cord lesions predict disease progression in radiologically isolated syndrome. Neurology. 2011 Feb 22;76(8):686-92. doi: 10.1212/WNL.0b013e31820d8b1d. Epub 2011 Jan 26. PMID 21270417
- [Result] Okuda DT, Mowry EM, Beheshtian A, Waubant E, Baranzini SE, Goodin DS, Hauser SL, Pelletier D. Incidental MRI anomalies suggestive of multiple sclerosis: the radiologically isolated syndrome. Neurology. 2009 Mar 3;72(9):800-5. doi: 10.1212/01.wnl.0000335764.14513.1a. Epub 2008 Dec 10. PMID 19073949
- [Derived] Okuda DT, Kantarci O, Lebrun-Frenay C, Sormani MP, Azevedo CJ, Bovis F, Hua LH, Amezcua L, Mowry EM, Hotermans C, Mendoza J, Walsh JS, von Hehn C, Vargas WS, Donlon S, Naismith RT, Okai A, Pardo G, Repovic P, Stuve O, Siva A, Pelletier D. Dimethyl Fumarate Delays Multiple Sclerosis in Radiologically Isolated Syndrome. Ann Neurol. 2023 Mar;93(3):604-614. doi: 10.1002/ana.26555. Epub 2022 Dec 10. PMID 36401339
- See also: Tecfidera USPI — http://www.accessdata.fda.gov/drugsatfda_docs/label/2013/204063lbl.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tecfidera | Placebo
Started | 44 | 43
Completed | 30 | 29
Not Completed | 14 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tecfidera | Placebo | Total
Number analyzed (Participants) | 44 | 43 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.57 (12.87) | 44.81 (13.88) | 44.18 (13.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 61
  Male | 13 | 13 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 40 | 38 | 78
  Black or African American | 2 | 3 | 5
  Other | 2 | 2 | 4
Expanded Disability Status Scale (EDSS) [Median (Full Range); unit: units on a scale] — The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
  units on a scale | 1 [0 to 3] | 1 [0 to 3] | 1 [0 to 3]
Multiple Sclerosis (MS) family history [Count of Participants; unit: Participants] | 3 | 6 | 9
Presence of gadolinium enhancing lesions [Count of Participants; unit: Participants] — Population: 11 missing data
  Participants
    number analyzed (Participants) | 38 | 38 | 76
    (all) | 6 | 2 | 8
T2-weighted hyperintense lesion volume [Mean (Standard Deviation); unit: mm^3] — Population: 4 missing data
  mm^3
    number analyzed (Participants) | 40 | 43 | 83
    (all) | 7.30 (1.07) | 7.32 (0.89) | 7.31 (0.97)

OUTCOME MEASURES:

1. Primary Outcome: The Time From Randomization to the First Demyelinating Event (Acute or Development of an Initial Symptom Resulting in a Progressive Clinical Course)
Description: The primary outcome measure for this trial is the time to the first acute or progressive neurological event resulting from CNS demyelination from randomization into the trial.
Time Frame: 96 weeks
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Tecfidera | Placebo
Number analyzed (Participants) | 44 | 43
weeks | 89.69 (23.99) | 77.81 (32.19)

2. Secondary Outcome: Change in Lesion Volume on T2-weighted MRI
Description: Change in lesion volume on T2-weighted MRI is measured by follow-up MRI at 96 weeks in the placebo group and in the Tecfidera group.
Time Frame: Baseline, 96 weeks
Population: 3 participants out of 30 who completed the assigned treatment, their baseline MRI data was missing and hence were not analyzed.
  3 participants out of 29 who completed the assigned placebo arm, their MRI data was not collected due to technical issues and hence were not analyzed.
Measure: Mean (Standard Deviation); unit: mm³
Arm/Group | Tecfidera | Placebo
Number analyzed (Participants) | 27 | 26
mm³ | 0.005 (0.03) | 0.04 (0.03)

3. Secondary Outcome: Number of Newly Enlarging T2 Lesions
Description: Number of newly enlarging T2 lesions is measured by follow-up MRI at 96 weeks in the placebo group and in the Tecfidera group.
Time Frame: 96 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T2 lesions
Arm/Group | Tecfidera | Placebo
Number analyzed (Participants) | 27 | 26
T2 lesions | 0.03 (0.003) | 0.10 (0.07)

4. Secondary Outcome: Number of New T2 Lesions
Description: Number of new T2 lesions as measured by follow-up MRI at 96 weeks in the placebo group and in the Tecfidera group.
Time Frame: 96 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T2 lesions
Arm/Group | Tecfidera | Placebo
Number analyzed (Participants) | 27 | 26
T2 lesions | 0.09 (0.06) | 0.54 (0.28)

5. Secondary Outcome: Newly Enlarging T2 Lesions and New T2 Lesions Combined
Description: Newly enlarging T2 lesions and new T2 lesions combined is measured by follow-up MRI at 96 weeks in the placebo group and in the Tecfidera group.
Time Frame: 96 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T2 lesions
Arm/Group | Tecfidera | Placebo
Number analyzed (Participants) | 27 | 26
T2 lesions | 0.12 (0.07) | 0.62 (0.30)

6. Secondary Outcome: Number of Contrast Enhancing Lesions
Description: Number of contrast enhancing lesions is measured by follow-up MRI at 96 weeks in the placebo group and in the Tecfidera group.
Time Frame: 96 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: contrast enhancing lesions
Arm/Group | Tecfidera | Placebo
Number analyzed (Participants) | 27 | 26
contrast enhancing lesions | 0.07 (0.38) | 0 (0)

7. Secondary Outcome: Change in the Number of Participants With Brain Atrophy
Description: Change in the number of participants with brain atrophy is measured by follow-up MRI at 96 weeks in the placebo group and in the Tecfidera group.
Time Frame: Baseline, 96 weeks
Population: Data were not collected.
Arm/Group | Tecfidera | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse Events (AE) occurred during 2 years of follow up. AEs were routinely determined through regular investigator assessment.
Arm/Group | Tecfidera | Placebo
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/43
Serious Adverse Events (participants affected / at risk) | 4/44 | 4/43
Other Adverse Events (participants affected / at risk) | 44/44 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tecfidera (N=44) | Placebo (N=43)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spondylolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Spontaneous cerebrospinal fluid leak syndrome (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tecfidera (N=44) | Placebo (N=43)
Vision blurred (Eye disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 1 (1)
Chest discomfort (General disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 4 (4) | 4 (4)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2)
Sinusitis (Infections and infestations) | 5 (6) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 3 (7) | 1 (1)
Blood glucose increased (Investigations) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 7 (8) | 6 (6)
Hypoaesthesia (Nervous system disorders) | 6 (6) | 5 (6)
Paraesthesia (Nervous system disorders) | 6 (6) | 5 (6)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Flushing (Vascular disorders) | 22 (24) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT02739542/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT02739542/SAP_001.pdf
  • Informed Consent Form (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT02739542/ICF_002.pdf